CLINICAL TRIAL: NCT01197846
Title: Efficacy of Quetiapine XR vs. Placebo as Concomitant Treatment to Mood Stabilizers in the Control of Subsyndromal Symptoms of Bipolar Disorder
Brief Title: Efficacy of Quetiapine XR Versus Placebo as Concomitant Treatment to Mood Stabilizers in the Control of Subsyndromal Symptoms of Bipolar Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centro de Investigación Biomédica en Red de Salud Mental (Network)
Responsible Party: Principal Investigator, Celso Arango Lopez, MD; PhD, Centro de Investigación Biomédica en Red de Salud Mental
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D1443L00079
Record Dates: First submitted 2010-09-02; First posted 2010-09-09 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quetiapine (Experimental): Quetiapine 300 mg or 600 mg
  Interventions: Drug: Quetiapine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Quetiapine — quetiapine 300 mg or 600 mg
  Other Names: Quetiapine XR
  Arms: Quetiapine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Pilot multicentric, prospective, placebo controlled, randomized double blinded, study of 12 weeks follow-up Adult patients diagnosed of bipolar disorder I or II, in previous treatment with no more than two concomitant mood stabilizers at stable doses and current subsyndromal symptoms, defined as YMRS ≤14 and/ or MADRS≥8 and ≤14 would be included Sub-acute phases would be excluded (at least 8 weeks from last exacerbation would be required for inclusion).

DETAILED DESCRIPTION:
Remission of acute episodes usually doesn't correlate with symptomatic or functional recovery in occupational and social domains after (McQueen et al, 2001; Tohen et al, 2000) Ongoing depressive symptoms are the strongest predictor of functional deficits in persons with bipolar disorder (Bauer et al, 2001; Judd et al, 2005). Depressive subsyndromal symptoms are associated to functional impairment in bipolar disorder (Vojta et al, 2001; Altshuler et al, 2002; Yatham et al, 2004) The addition of olanzapine to valproate or lithium provided superior efficacy to valproate or lithium plus placebo in non completely remitted manic and mixed bipolar episodes, mainly through a control of depressive symptoms (Tohen et al, 2002) Quetiapine has demonstrated to be efficacious in the control of depressive symptoms in Bipolar Disorder (BOLDER, EMBOLDEN studies) and in the prevention of recurrences, maintaining the patient in YMRS and MADRS scores under the cut-off point between asymptomatic and subsyndromal states (Studies 126, 127 and 144) Thus it's expectable that adding quetiapine to previous mood stabilizers in bipolar patients with subsyndromal symptoms probably would improve their symptoms, mainly depressive, to levels not only of syndromic but of symptomatic remission, driving to a better functional status Quetiapine extended release would be used because its advantages on quetiapine immediate release regarding an easier and comfortable posology and potential better adherence

ELIGIBILITY:
Inclusion Criteria:

1. Informed Consent signature
2. At least 18 years old
3. Diagnoses of bipolar disorder I or II (as DSM-IV-TR 4ª Ed codes)
4. Previous treatment with a mood stabilizer (lithium, valproate or lamotrigine) at stable and optimum doses for at least six weeks prior to the start of the trial (i.e., on the same dose and serum levels within the therapeutic ranges: 0.6-1.2 mEq/l of lithium or 50-100 ug/ml of valproate)
5. Presenting subsyndromal symptoms at enrolment and randomization point, defined as YMRS ≤ 14 and/ or MADRS ≥ 8 and ≤14
6. At least one manic, mixed, or depressed episode in the last 5 years
7. Being able to understand and meet the study requirements

Exclusion Criteria:

1. Pregnant or nursing women
2. Mental retardation.
3. Current active diagnoses of any axis I or II DSM-IV-TR diagnoses different from bipolar disorder I or II. This doesn't apply to nicotine nor caffeine abuse-dependence. Punctual alcohol and/or substances use not constitutive of a diagnoses of abuse or dependence following DSM-IV-TR criteria wouldn't suppose the exclusion of the patient from the study. Anxiety in levels not constitutive of any anxiety disorder within those codified in DSM-IV-TR wouldn't either suppose the exclusion of the patient from the study
4. Having suffered any acute episode (depressive, manic, or mixed) within the 8 weeks prior to enrolment, as defined in DSM-IV-TR
5. Patients that, in the investigator's opinion, are at a high risk of suicide or mean a risk of aggression to others.
6. Having been treated with any antidepressant at randomization.
7. Having been treated with any mood stabilizer other than lithium/valproate/lamotrigine at randomization.
8. Having been treated with any oral antipsychotic drug at randomization. Administration of a depot antipsychotic medication within one dosing interval prior to randomization (e.g. Long acting Risperidone 2 weeks; Zuclopenthixol 4 weeks; Pipotiazine 4 weeks; Flufenazine 6 weeks)
9. Having been treated with any of the following P450-3A4 cytochrome inhibitors in the 14 days prior to inclusion, including: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, fluvoxamine, indinavir, nelfinavir, ritonavir and saquinavir.
10. Having been treated with any of the following P450-3A4 cytochrome inducers in the 14 days prior to inclusion, including: phenytoin, carbamazepine, barbiturates, rifampicin, St. John's wart, and glucocorticoids.
11. Any contraindication to the use of quetiapine fumarate in the investigator's opinion (including lack of response to it in previous treatment attempts)
12. Suffering any medical condition that can effect the absorption, distribution, metabolism or excretion of the study treatment(s).
13. Suffering any medical condition in decompensation or not receiving inappropriate treatment for it in the investigator's opinion (e.g., hyperthyroidism, angina pectoris, hypertension...)
14. Suffering unstable diabetes at enrolment or randomization
15. Absolute neutrophil count ≤ 1.5 x 109 per litre at randomization
16. Non-compliance with the study plan.
17. Participation in another clinical trial in the four weeks prior to randomization

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-09; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
To assess the efficacy of quetiapine extended release (QTP XR) vs. placebo in the control of bipolar subsyndromal symptoms when added to previous mood stabilizer treatment (lithium/ valproate/lamotrigine) | Study of 12 weeks follow-up

SECONDARY OUTCOMES:
To assess the efficacy of QTP XR vs. placebo when added to previous mood stabilizer treatment (lithium/ valproate/lamotrigine) in functional level of bipolar patients with subsyndromal symptoms | Study of 12 weeks follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Vieta, PhD, Principal Investigator — Hospital Clinic I Provincial. Barcelona. Spain; Ana Gonzalez Pinto, Principal Investigator — Hospital Santiago Apostol. Vitoria. Spain; Benedikt Amann, Principal Investigator — Hospital Benito Menni. Barcelona. Spain; Celso Arango, Principal Investigator — Hospital General Universitario Gregorio Marañon. Madrid. Spain; Jose Manuel Crespo, Principal Investigator — Hospital Universitari de Bellvitge. Barcelona. Spain; Julio Bobes, Principal Investigator — Centro de Salud Mental II. Oviedo. Spain; Josefina Perez, Principal Investigator — Hospital Santa Creu I Sant Pau. Barcelona. Spain; Gabriel Selva, Principal Investigator — Hospital Clinico de Valencia/ CSM Foios. Valencia. Spain; Belen Arranz, Principal Investigator — Parc Sanitari Sant Joan de Deu. Barcelona. Spain; Jeronimo Saiz, Principal Investigator — Hospital Universitario Ramon y Cajal. Madrid. Spain
Locations (10):
- Spain (10):
  - Hospital Santa Creu I Sant Pau, Barcelona, Barcelona
  - Hospital Clinic I Provincial, Barcelona, Barcelona
  - Hosptial Benito Menni, Barcelona, Barcelona
  - Hospital Universitari de Bellvitge, Barcelona, Barcelona
  - Parc Sanitari Sant Joan de Deu, Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid
  - Hospital Universitario Ramon Y Cajal, Madrid, Madrid
  - Centro de Salud Menta II, Oviedo, Oviedo
  - Hosptial Clinico Valencia/ CSM Foios, Valencia, Valencia
  - Hospital Santiago Apostol, Vitoria-Gasteiz, Vitoria